CLINICAL TRIAL: NCT01358708
Title: Treatment of Diarrhea-predominant Irritable Bowel Syndrome With LACTEOL® 340 mg: A Pilot Study Evaluating Safety and Efficacy
Brief Title: Treatment of Diarrhea-predominant Irritable Bowel Syndrome (IBS-D) With LACTEOL® 340 mg
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MA-LA-IBS09-01
Record Dates: First submitted 2010-05-16; First posted 2011-05-24 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Diarrhea-predominant Irritable Bowel Syndrome
MeSH Terms: interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LACTEOL® 340 mg (Experimental)
  Interventions: Drug: LACTEOL® 340 mg
- PLACEBO (Placebo Comparator)
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: LACTEOL® 340 mg — LACTEOL® 340 mg will be taken for a 4-week duration (28 days) as three capsules a day: two capsules in the morning and one capsule in the evening.
  Arms: LACTEOL® 340 mg
Drug: PLACEBO — Matched LACTEOL® 340 mg Placebo will be taken for a 4-week duration (28 days) as three capsules a day: two capsules in the morning and one capsule in the evening.
  Arms: PLACEBO

SUMMARY:
Irritable bowel syndrome is a complex condition with a high unmet medical need for effective and safe treatment options. Lacteol® is a lactobacillus product used for adjunctive and symptomatic treatment of diarrhea. In this study, Lacteol® 340 mg will be evaluated as a potential therapy for the treatment of diarrhea-predominant irritable bowel syndrome (IBS-D).

DETAILED DESCRIPTION:
This study will include the following phases: Screening Phase, Run-In Phase, Double-Blind Treatment Phase and Open-Label Treatment Phase.

Screening: Eligibility of subjects will be evaluated following informed consent signature. Screening procedures/evaluations (physical exam, concomitant medications, clinical laboratory tests) and confirmation of eligibility following Rome III Diagnostic questionnaire will be performed.

Run-In: Subjects will enter a 2-week Run-In Phase during which IBS Symptoms and Stool Characteristics will be recorded. At the end of the Run-In Phase, data collected over the last week will be reviewed. Upon confirmation of IBS-D severity status, subjects may be randomized.

Double-Blind Treatment: Subjects will take study medication (either LACTEOL® 340 mg or Placebo) for 28 days. During this time, IBS Symptoms and Stool Characteristics and global assessment of relief will be recorded, and clinical laboratory tests will be performed. HAD score will be assessed at the end of the double blind treatment.

Open-Label Treatment: All study completers will be eligible for a second 28 day Open-Label Treatment in the event that IBS-D symptoms remain or recur within the month following the end of Double-Blind Treatment. Subjects will take the study medication (LACTEOL® 340 mg) for 28 days. During this time, IBS Symptoms and Stool Characteristics and global assessment of relief will be recorded, and clinical laboratory tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

* IBS-D diagnosis using the Rome III questionnaire
* IBS Symptoms Severity Scale (IBS-SSS) score ranging between 100 and 400
* Bristol Stool Form Scale score exceeding two (> 2) but less than seven (< 7)
* Stable diet
* Mental and legal ability to sign informed consent

Exclusion Criteria:

* Diagnosis of Inflammatory Bowel Disease (IBD)
* Chronic use of systemic steroids
* Diagnosis of autoimmune Diseases or Disorders
* Invasive abdominal surgery
* Use of antibiotics prior to screening
* Allergy to active substance or any other ingredient in LACTEOL® 340 mg
* Congenital galactosemia, glucose, fructose and/or galactose malabsorption syndrome, lactase deficiency or lactose intolerance
* Diagnosis of exocrine pancreatic insufficiency
* Use of any experimental drug within the 30 days prior to screening

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan T Shaw, PhD, Study Director — Axcan Pharma Inc.
Locations (8):
- France (5):
  - Bordeaux
  - Colombes
  - Marseille
  - Nice
  - Rouen
- Germany (3):
  - Berlin
  - Hamburg
  - Mannheim

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject in: 22 June 2010; last subject out: 12 September 2011; ten (10) sites were recruited to participate in this trial and 7 of these (4 in France and 3 in Germany) enrolled subjects.
Pre-assignment Details: Inclusion criteria related to symptom severity and stool characteristics assessed during 2nd week of Run-In Phase; ≥ 5 days of symptom data necessary for randomization; Double-Blind Phase completers eligible for a 28-day open-label treatment with LACTEOL® if symptoms not improved or recurring within 1 month after end of blinded treatment.
Groups:
- LACTEOL® 340 mg: LACTEOL® active medication was taken for a 4-week duration (28 days) as three capsules a day: two capsules in the morning and one capsule in the evening.
- PLACEBO: Matched LACTEOL® placebo was taken for a 4-week duration (28 days) as three capsules a day: two capsules in the morning and one capsule in the evening.
Period: Double-Blind Treatment Phase
Arm/Group | LACTEOL® 340 mg | PLACEBO
Started | 13 | 13
Randomized | 13 | 13
Received Study Medication | 12 (For 1 subject, unused med not returned to the site and intake of study medication not confirmed.) | 13
Completed | 10 | 13
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 0
Period: Open-Label Treatment Phase
Arm/Group | LACTEOL® 340 mg | PLACEBO
Started | 5 (Number of subjects on LACTEOL® during double-blind treatment and entering the Open-Label Phase) | 12 (Number of subjects on PLACEBO during double-blind treatment and entering the Open-Label Phase)
Completed | 5 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis conducted on the Intent-to-Treat population defined as all randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | LACTEOL® 340 mg | PLACEBO | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  France | 6 | 6 | 12
  Germany | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Global Assessment of Relief During the Double-Blind Treatment Phase Using the Subject Global Assessment (SGA)
Description: Subjects were considered as responders if they had answered "Yes" to the following question at least 50% of the time during the 4-week treatment phase: "Over the past week, do you consider that you have had satisfactory relief from your IBS symptoms?"
Time Frame: Weekly Assessment (every 7 days)
Population: Analysis conducted on the Intent-to-Treat population defined as all randomized subjects; observed case (OC) data with no imputation made
Measure: Number; unit: percentage of participants
Arm/Group | LACTEOL® 340 mg | PLACEBO
Number analyzed (Participants) | 13 | 13
percentage of participants
  Responders | 30.8 | 30.8
  Non-responders | 69.2 | 69.2

2. Secondary Outcome: Global Assessment of Relief During the Open-Label Treatment Phase Using the Subject Global Assessment (SGA)
Description: as for outcome 1
Time Frame: Weekly Assessment (every 7 days)
Population: Analysis conducted on the Intent-to-Treat population defined as all subjects randomized to double-blind treatment and who subsequently entered the Open-Label Treatment Phase; observed case (OC) data with no imputation made; SGA data not available for one patient so that the analysis was performed on 16 rather than 17 patients
Measure: Number; unit: percentage of participants
Arm/Group | LACTEOL® 340 mg
Number analyzed (Participants) | 16
percentage of participants
  Responders | 50.0
  Non-responders | 50.0

3. Secondary Outcome: Symptom Severity During the Double-Blind Treatment Phase Using the IBS Symptom Severity Scale (IBS-SSS) Total Score
Description: The IBS-SSS has five questions related to four domains: abdominal pain severity and duration, abdominal distension, dissatisfaction with bowel habit and quality of life. The IBS-SSS score ranges from 0 (best outcome) to 500 (worst outcome).
Time Frame: Weekly assessment (every 7 days)
Population: Analysis conducted on the Intent-to-Treat population defined as all randomized subjects; observed case (OC) data with no imputation made. Number of participants analyzed refers to number of participants at Baseline.
Measure: Mean (Standard Deviation); unit: units on a scale (from 0 to 500)
Arm/Group | LACTEOL® 340 mg | PLACEBO
Number analyzed (Participants) | 13 | 13
units on a scale (from 0 to 500)
  Baseline IBS-SSS score | 245.0 (87.3) | 307.5 (72.36)
  IBS-SSS score at end of Week 1 (Day 7) | 219.2 (76.36) | 271.2 (109.72)
  IBS-SSS score at end of Week 2 (Day 14) | 229.5 (81.95) | 265.4 (99.93)
  IBS-SSS score at end of Week 3 (Day 21) | 233.6 (87.78) | 254.8 (103.75)
  IBS-SSS score at end of Week 4 (Day 28) | 228.6 (91.82) | 241.4 (99.23)

4. Secondary Outcome: Stool Characteristics During the Double-Blind Treatment Phase Using the Bristol Stool Form Scale
Description: The Bristol Stool Form Scale score ranges from 1 to 7 from hard (score of 1) to watery (score of 7). Data are presented as the mean of daily assessments over a week.
Time Frame: Daily assessment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale (from 1 ato 7)
Arm/Group | LACTEOL® 340 mg | PLACEBO
Number analyzed (Participants) | 13 | 13
units on a scale (from 1 ato 7)
  Baseline Bristol Stool Form Scale Score | 4.8 (1.14) | 4.9 (0.64)
  Bristol Stool Form Score during Week 1 | 4.3 (1.29) | 4.8 (0.61)
  Bristol Stool Form Score during Week 2 | 4.6 (1.33) | 4.8 (0.83)
  Bristol Stool Form Score during Week 3 | 4.4 (1.52) | 4.4 (0.78)
  Bristol Stool Form Score during Week 4 | 4.4 (1.32) | 4.8 (0.81)

5. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Score During the Double-Blind Phase
Description: The HADS has 14 questions related to 2 domains: Anxiety subscale (7 questions) and Depression subscale (7 questions). Each question is graded from 0 (best outcome) to 3 (worst outcome), for a total score ranging from 0 (best outcome) to 42 (worst outcome).
Time Frame: At Screening and End of Double-Blind Treatment Phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale (from 0 to 42)
Arm/Group | LACTEOL® 340 mg | PLACEBO
Number analyzed (Participants) | 13 | 13
units on a scale (from 0 to 42)
  Baseline HADS Total Score | 9.7 (5.14) | 10.7 (4.82)
  HADS Total Score at End of Double-Blind Treatment | 9.9 (6.10) | 9.5 (5.88)

6. Secondary Outcome: Symptom Severity During the Open-Label Treatment Phase Using the IBS Symptom Severity Scale (IBS-SSS) Total Score
Description: as for outcome 3
Time Frame: Weekly assessment (every 7 days)
Population: Analysis conducted on the Intent-to-Treat population defined as all subjects randomized to double-blind treatment and who subsequently entered the Open-Label Treatment Phase; observed case (OC) data with no imputation made; baseline defined as the last non-missing assessment prior to the first dose of double-blind medication.
Measure: Mean (Standard Deviation); unit: units on a scale (from 0 to 500)
Arm/Group | LACTEOL® 340 mg
Number analyzed (Participants) | 17
units on a scale (from 0 to 500)
  Double-Blind Baseline IBS-SSS score | 270.5 (78.2)
  IBS-SSS score at end of Week 1 (Day 7) | 224.6 (73.06)
  IBS-SSS score at end of Week 2 (Day 14) | 211.5 (93.58)
  IBS-SSS score at end of Week 3 (Day 21) | 199.2 (103.68)
  IBS-SSS score at end of Week 4 (Day 28) | 222.5 (103.14)

7. Secondary Outcome: Stool Characteristics During the Open-Label Treatment Phase Using the BSFS
Description: The Bristol Stool Form Scale (BSFS) score ranges from 1 to 7 from hard (score of 1) to watery (score of 7). Data are presented as the mean of daily assessments over a week.
Time Frame: Daily assessment
Population: Analysis conducted on the Intent-to-Treat population defined as all subjects randomized to double-blind treatment and who subsequently entered the Open-Label Treatment Phase ; observed case (OC) data with no imputation made; baseline defined as the last non-missing assessment prior to the first dose of double-blind study medication
Measure: Mean (Standard Deviation); unit: units on a scale (from 1 to 7)
Arm/Group | LACTEOL® 340 mg
Number analyzed (Participants) | 17
units on a scale (from 1 to 7)
  Double-Blind Baseline BSFS Score | 5.0 (0.68)
  BSFS score during Week 1 | 4.6 (1.10)
  BSFS score during Week 2 | 4.5 (1.24)
  BSFS score during Week 3 | 4.4 (1.45)
  BSFS score during Week 4 | 4.4 (1.33)

8. Secondary Outcome: Use of Rescue Medication During the Double-Blind and Open-Label Treatment Phases of the Study
Description: Number of subjects using rescue medication (bisacodyl or loperamide) during each treatment phase of the study
Time Frame: 8 weeks
Population: Analysis conducted on the Intent-to-Treat population for both treatment phases
Measure: Number; unit: participants
Groups:
- LACTEOL® 340 mg Double-Blind Period; LACTEOL® 340 mg Open-Label Period: LACTEOL® active medication was taken for a 4-week duration (28 days) as three capsules a day: two capsules in the morning and one capsule in the evening.
- PLACEBO Double-Blind Period: Matched LACTEOL® placebo was taken for a 4-week duration (28 days) as three capsules a day: two capsules in the morning and one capsule in the evening.
Arm/Group | LACTEOL® 340 mg Double-Blind Period | PLACEBO Double-Blind Period | LACTEOL® 340 mg Open-Label Period
Number analyzed (Participants) | 13 | 13 | 17
participants | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Informed Consent Form signature up to 28 days following the end of double-blind treatment (symptom recurrence observation period) or up to End of Open-Label Treatment Phase Visit (Days 29 to 38) for subjects continuing with open-label treatment
Description: Adverse events collected during study visits as well as via an interactive voice response system (IVRS) while at home; clinical labs performed at baseline and end of each period; only treatment-emergent adverse events are displayed, ie. events that occurred or worsened in intensity on or after the first dose of study medication in each period.
Arm/Group | LACTEOL® 340 mg Double-Blind Period | PLACEBO Double-Blind Period | LACTEOL® 340 mg Open-Label Period
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/17
Other Adverse Events (participants affected / at risk) | 2/13 | 2/13 | 2/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LACTEOL® 340 mg Double-Blind Period (N=13) | PLACEBO Double-Blind Period (N=13) | LACTEOL® 340 mg Open-Label Period (N=17)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Because of early termination of this trial, the number of subjects analyzed was too small to perform statistical analyses and draw conclusions relative to the efficacy and safety of LACTEOL®.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions vary in accordance with each agreement with the individual investigators. Sponsor will allow publication after a multi-center publication has been published or after an agreed period of time if no such multi-center publication is submitted for publication. Sponsor can ask that Sponsor's confidential information be removed from any publication and can defer publication for a period of time to allow for Sponsor to obtain patent or other intellectual property right protection.